CLINICAL TRIAL: NCT05572034
Title: Cardiac Autonomic Denervation for Cardio-inhibitory Syncope
Acronym: CardioSync
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Abbott (Industry)
Responsible Party: Principal Investigator, Mauricio Ibrahim Scanavacca, Director of arrhythmia and electrophysiology Unit, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UAP 174
Record Dates: First submitted 2022-05-20; First posted 2022-10-07 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Bradycardia; Syncope; Syncope, Vasovagal
Keywords: Cardiac denervation; Cardio-inhibitory syncope
MeSH Terms: conditions — Bradycardia; Syncope; Syncope, Vasovagal

STUDY DESIGN:
Intervention Model Description: randomized, prospective, sham controll, on a 1:1:1 basis to group A (Sham - 15 patients); group B (right sided denervation - 15 patients); and group C (bilateral denervation - 15 patients)
Who Masked: Participant
Masking Description: all patients will go for intervention, however they will not know which group they were randomized to
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Sham Comparator): A diagnostic electrophysiological study will be performed in patients of group A
  Interventions: Procedure: Electrophysiological study
- Group B (Active Comparator): A electrophysiological study with cardiac denervation, with right Ganglionated Plexi ablation exclusively will be performed in patients of group B
  Interventions: Procedure: Electrophysiological study and Right side Ganglionated Plexi ablation
- Group C (Active Comparator): A electrophysiological study with cardiac denervation, with right and left Ganglionated Plexi ablation will be performed in patients of group C.
  Interventions: Procedure: Electrophysiological study and bi-atrial Ganglionated Plexi ablation

INTERVENTIONS:
Procedure: Electrophysiological study — Electrophysiological study: patients in a fasting state and under total intravenous anesthesia Intracardiacelectrogramsare displayed simultaneously on a multichannel recorder. Programmed atrial and ventricular stimulation are performed to rule out sustained arrhythmias, primary conduction system dysfunction, and sick sinus syndrome.
  Arms: Group A
Procedure: Electrophysiological study and Right side Ganglionated Plexi ablation — Electrophysiological study: patients in a fasting state and under total intravenous anesthesia Intracardiacelectrogramsare displayed simultaneously on a multichannel recorder. Programmed atrial and ventricular stimulation are performed to rule out sustained arrhythmias, primary conduction system dysfunction, and sick sinus syndrome.
  GP Mapping and Cardiac denervation: Specific atrium sites are empirically identified as GP by presumed anatomic location based on previous works (anatomic mapping):
  In the RA: the posterior aspect of the interatrial septum, between the posterior wall and coronary sinus ostium; and, the septal aspect of the superior vena cava junction (opposite to the LA GP tags).
  A 3.5-mm irrigated tip catheter will be used to deliver radiofrequency energy (50°C, 20-30 W, for 30-60 seconds) with a 17 mL/min irrigation flow.
  Arms: Group B
Procedure: Electrophysiological study and bi-atrial Ganglionated Plexi ablation — Electrophysiological study: patients in a fasting state and under total intravenous anesthesia Intracardiacelectrogramsare displayed simultaneously on a multichannel recorder. Programmed atrial and ventricular stimulation are performed to rule out sustained arrhythmias, primary conduction system dysfunction, and sick sinus syndrome.
  GP Mapping and Cardiac denervation: Specific atrium sites are empirically identified as GP by presumed anatomic location based on previous works(anatomic mapping):
  In the LA: the inferior right GP (septal aspect of the right pulmonary veins [PV]) antra, and LA posterior wall. In the RA: the posterior aspect of the interatrial septum, between the posterior wall and coronary sinus ostium; and the septal aspect of the superior vena cava junction (opposite to the LA GP tags).
  A 3.5-mm irrigated tip catheter will be used to deliver radiofrequency energy (50°C, 20-30 W, for 30-60 seconds) with a 17 mL/min irrigation flow.
  Arms: Group C

SUMMARY:
Background: Autonomic system modification is an established therapeutic approach that has been increasingly used for the treatment of vagal-related symptomatic bradycardia, such as cardio-inhibitory vasovagal syncope1-12.

Although convincing results had been reported from small populations, a large randomized study providing robust evidence on the efficacy of this approach has not yet been performed.

Hypothesis: Cardiac autonomic system modification is effective for the treatment of vagal-related symptomatic bradycardia, and is associated better clinical results as compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 70 years old.
* Cardio-inhibitory response (VASIS 2A or 2B) during tilt test, or after carotid sinus massage.
* Patients with bradycardia mediated by vagal hypertonia documented on 24-hour Holter monitoring and a clear relationship with symptoms.

Exclusion Criteria:

* Ages under 18 and over 70
* Presence of structural heart disease documented by echocardiography.
* Hypothyroidism and hyperthyroidism, drug effects, obstructive sleep apnea and other causes of secondary bradycardia.
* Anatomical disease of the conduction system.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
recurrence of syncope | 24 months
  To compare the recurrence of syncope or pre-syncope and a negative tilt test with the different techniques of electrophysiological procedures currently used.

SECONDARY OUTCOMES:
electrocardiographic and electrophysiological parameters | 24 months
  Compare the following electrocardiographic and electrophysiological parameters of vagal attenuation:
  * Heart rate (bpm - beats per minute);
  * Internal AH (represents AV internodal conduction time, with normal values between 50-120 ms);
  * Wenckebach cycle;
  * Presence of Holter pauses 30 days after the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Mauricio I Scanavacca, MD, PhD, Principal Investigator — University of Sao Paulo - General Hospítal
Locations (2):
- Brazil (2):
  - University of Sao Paulo General Hospital, São Paulo, São Paulo
  - Arrhythmia and electrophysiology of the Heart Institute - University of São Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hardy C, Rivarola E, Scanavacca M. Role of Ganglionated Plexus Ablation in Atrial Fibrillation on the Basis of Supporting Evidence. J Atr Fibrillation. 2020 Jun 30;13(1):2405. doi: 10.4022/jafib.2405. eCollection 2020 Jun-Jul. PMID 33024505
- [Background] Sarabanda AV, Melo SL, Rivarola E, Hachul D, Scanavacca M. Anatomically guided atrial ganglionated plexus ablation evaluated by extracardiac vagal stimulation for vagally mediated atrioventricular block. HeartRhythm Case Rep. 2021 Feb 10;7(5):301-305. doi: 10.1016/j.hrcr.2021.02.002. eCollection 2021 May. No abstract available. PMID 34026520